CLINICAL TRIAL: NCT06813443
Title: Clinical, Instrumental, and Molecular (Circulating and Tissue microRNAs) Characterization of Patients With Cardiomyopathy to Identify Critical Patients With Severe Organ Failure to be Candidates for Cardiac Transplantation
Brief Title: Characterization of Patients With Cardiomyopathy to Identify Critical Patients Candidates for Cardiac Transplantation
Acronym: CMPMIRNA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CMPMIRNA; RC-2022-277327/RC-2024-2789983 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2025-01-09; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-12

CONDITIONS: Cardiomyopathies; Amyloidosis Cardiac; Fabry Disease; Arrhythmogenic Cardiomyopathy; Hypertrophic Cardiomyopathy (HCM); Laminopathies; Dystrophia Myotonica; Mitochondrial Cardiomyopathy; Dilated Cardiomyopathy; Sudden Cardiac Death; Heart Transplantation; Glycogen Storage Disease; Infiltrative Cardiomyopathy; Cardiac Magnetic Resonance Imaging; Electrocardiogram; Micro RNA; Echocardiogram
Keywords: cardiomyopathy; cardiac amyloidosis; Fabry disease; hypertrophic cardiomyopathy; dilated cardiomyopathy; sudden cardiac death; arrhythmogenic cardiomyopathy; heart failure; heart transplantation
MeSH Terms: conditions — Cardiomyopathies; Amyloid Neuropathies, Familial; Fabry Disease; Cardiomyopathy, Hypertrophic; Laminopathies; Myotonic Dystrophy; Cardiomyopathy, Dilated; Death, Sudden, Cardiac; Glycogen Storage Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to identify new diagnostic and prognostic markers for CMP that can help predict disease progression. In particular, the study will focus on microRNAs (miRNAs) and spatial transcriptomics, which are emerging techniques that may provide insights into the underlying disease mechanisms. By understanding these markers, the investigators hope to improve the way the investigators diagnose and manage CMP, particularly in terms of predicting progression to heart failure or heart transplantation.

The study will evaluate patients with hypertrophic cardiomyopathy (e.g., sarcomeric forms, Anderson-Fabry disease, AL, and TTR cardiac amyloidosis), dilated cardiomyopathy and arrhythmogenic cardiomyopathy. These patients will undergo clinical evaluations, including ECG, echocardiograms, CMR, biopsy analysis, and genetic testing, as well as molecular studies such as transcriptomics and miRNA analysis. This comprehensive approach aims to identify potential new biomarkers for diagnosing and predicting the disease course.

DETAILED DESCRIPTION:
This is a non-pharmacological, national multicenter cohort study with both retrospective and prospective components.

For the prospective study, patients with CMP will be consecutively enrolled from the outpatient or inpatient settings of the IRCCS Azienda Ospedaliero-Universitaria di Bologna (coordinating center), Azienda Ospedaliero-Universitaria Careggi di Firenze, and the Department of Cardiothoracic and Vascular Sciences, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome. Enrollment will begin upon receipt of favorable opinions from the respective Ethics Committees and general management approvals at each center until the planned sample size is reached.

For the retrospective study, all patients managed at the aforementioned centers prior to obtaining Ethics Committee approval and general management clearance will be included.

The structured collection of the data necessary for the evaluation of the objectives will be carried out by creating a specific electronic database in which retrospective data will be collected starting from January 1, 1990, and for the prospective observation period from the moment of ethical committee approval and receipt of the clearance from the general director until December 31, 2027. The electronic archive may be used to obtain or confirm new scientific evidence in the field of CMP, particularly with reference to diagnosis, prognosis, and therapy. The electronic archive will be compiled through the consultation of the clinical records (outpatient or hospitalization), from which data regarding demographics, remote and recent medical history, family history, any genetic investigations, instrumental tests, information about symptoms at onset, and therapy will be collected. Aside from the analysis of miRNAs on tissues, which will be carried out for the study and will not in any way affect the patients' diagnostic-therapeutic path, all instrumental exams and therapies that patients will undergo are part of standard clinical practice. Any genetic investigations that patients may undergo are part of the regular care pathway and will be performed when clinically indicated, or if a precise etiological diagnosis is necessary, with consequent therapeutic implications, in the differential diagnosis between various forms of CMP, and when, in the context of familial forms, it may be useful for family screening. Patients will be enrolled during hospitalization or at the outpatient visit. After obtaining informed consent, patients will be evaluated based on clinical needs. There is no minimum duration for following the patient. In a subgroup of patients enrolled in the prospective study, additional molecular evaluations will be carried out on plasma and cardiac tissue. The blood sample-taken as per clinical practice-will be processed within 4 hours through centrifugation. After isolation, the plasma will be divided into aliquots of 500 µL and stored at -80°C. In the subpopulation of the study undergoing endomyocardial biopsy (diagnostic) or cardiac surgery (e.g., myectomy, valve replacement, etc.), according to the standard-of-care, fresh cardiac tissue will be collected. The cardiac tissue (taken during endomyocardial biopsy/cardiac surgery performed according to clinical practice) will be partially immersed in formalin and sent, as per normal procedure, to pathology where it will be processed for paraffin embedding, and a small fragment will be frozen and immediately embedded in OCT (optimal cutting temperature) and stored at -80°C. RNA will then be extracted and analyzed using NGS (next-generation sequencing) of small RNA, ddPCR (droplet digital Polymerase Chain Reaction), and spatial transcriptomics.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with CMP according to current international guidelines
* Age ≥ 12 years at the time of diagnosis
* Obtaining informed consent from the patient and the parent or legal guardian (in the case of patients aged < 18 years)

Exclusion Criteria:

* none

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study plans to enroll a population of 700 patients affected by CMP evaluated both in the inpatient and outpatient regime, at
  * IRCCS AOUBO (n=520)
  * Azienda Ospedaliero-Universitaria Careggi of Florence (n=90)
  * Department of Thoracic Cardiovascular Sciences, Fondazione Policlinico Universitario A. Gemelli IRCSS of Rome (n=90)
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
risk stratification | Enrollment in the prospective phase and collection of data for the retrospective phase: 30 months; Follow-up: 2 years, Data analysis: 6 months
  Accuracy of clinical, instrumental, histological, and molecular variables in identifying critical CMP patients or those at risk of organ transplantation. For each marker and their combinations, specificity, sensitivity, and AUC will be assessed.
  Unit of Measurement: sensitivity, specificity, and Area Under the Curve (AUC)

SECONDARY OUTCOMES:
Gene expression profile (transcriptomics) and microRNA analysis | Enrollment in the prospective phase: 30 months, Follow-up: 2 years, Data analysis: 6 months
  The tissues analyzed will consist of blood (plasma microRNA) and cardiac tissue (MicroRNA Quantification and Spatial Transcriptomics) on endomyocardial biopsy/cardiac surgery samples performed for diagnostic/therapeutic purposes.
  These analysis will allow us to evaluate transcripts specific to each cell and/or small groups of cells by mapping their location within the tissue organization. Gene expression data will be explored in association with the tissue images using dedicated analysis software
  Unit of Measurement: number of miRNA copies/µL
AL (Light Chain Amyloidosis) vs TTR (Transthyretin) differential diagnosis in cardiac amyloidosis | Enrollment: 30 months; Data analysis: 6 months
  Development of a diagnostic model integrating clinical (NYHA class), instrumental (left ventricle mass in g/m², BNP in pg/mL, Troponin in ng/dL), and molecular (miRNA copies/µL) variables to differentiate AL vs TTR cardiac amyloidosis.
  Unit of Measurement: sensitivity, specificity, and Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Biagini, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria
Locations (3):
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Emilia-Romagna/Bologna
  - Dipartimento di Scienze Toraciche Cardiovascolari, Fondazione Policlinico Universitario A. Gemelli IRCSS di Roma, Roma, Lazio/Roma
  - Azienda Ospedaliero-Universitaria Careggi di Firenze, Florence, Toscana/Firenze